CLINICAL TRIAL: NCT06438835
Title: Development & Evaluation of Pneumatic Artificial Muscle(PAM) for Patients With Ankle Foot Orthosis(AFO)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/703
Record Dates: First submitted 2024-05-03; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PneuFlex AFO Assist (Experimental)
  Interventions: Diagnostic Test: PneuFlex AFO Assist

INTERVENTIONS:
Diagnostic Test: PneuFlex AFO Assist — It features a pneumatic artificial muscle designed to enhance ankle foot orthosis functionally for patients with mobility issues.

SUMMARY:
Pneumatic Artificial Muscles (PAMs), inspired by the structure and function of natural muscles, offer a lightweight and adaptable solution compared to traditional rigid Ankle Foot Orthosis(AFOs).

DETAILED DESCRIPTION:
The development process involves design optimization to ensure proper, fit, functionality and durability. Researchers utilize advanced materials and manufacturing techniques to create PAMs that mimic the natural movement of the ankle joint while providing sufficient support and flexibility. Evaluation of PAMs involves rigorous testing in both laboratory settings and real world environments. Bio-mechanical analysis assesses the performance of PAMs during various activities such as walking, running and stair negotiation. Critical trails involving patients with AFOs provide valueable feedback on usability, comfort and overall satisfaction. Additionally, long-term studied monitor the durability and reliability of PAMs over extended periods of use. Overall, the development and evaluation of PAMs for patient with AFOs represent a significant advancement in assistive technology. By offering a more natural and adaptive solution for gait assistance, PAMs enhance mobility, independence and quality of life for individuals with mobility impairments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of droop foot
* Ability to tolerate pneumatic pressure
* Sufficient muscle strength activation

Exclusion Criteria:

* Allergy to materials used in device fabrication
* Severe muscle weakness preventing activation
* Uncontrolled hypertension, pregnancy.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Functional Mobility | 12 months
  Functional mobility is a person's physiological ability to move independently and safely in a variety of environments in order to accomplish functional activities or tasks and to participate in the activities of daily living, at home, work and in the community
Range of motion (ROM) | 12 months
  Range of motion means the extent or limit to which a part of the body can be moved around a joint or a fixed point; the totality of movement a joint is capable of doing. Range of motion of a joint is gauged during passive ROM (assisted) PROM or active ROM (independent) AROM.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Ghani rehabilitation centre. Opposite to Misaq-ul-mall, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No